CLINICAL TRIAL: NCT03150459
Title: Safety and Tolerability of the Combination of Simvastatin Plus Rifaximin in Patients With Decompensated Cirrhosis: a Multicenter, Double-blind, Placebo Controlled Randomized Clinical Trial.
Brief Title: Simvastatin Plus Rifaximin in Decompensated Cirrhosis
Acronym: LIVERHOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Judit Pich (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager. CTU Clínic, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIVERHOPE_SAFETY; 2016-004499-23 (EudraCT Number)
Record Dates: First submitted 2017-05-03; First posted 2017-05-12 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Cirrhoses, Liver
MeSH Terms: interventions — Simvastatin; Rifaximin

STUDY DESIGN:
Intervention Model Description: Phase II, multicenter, double-blind placebo controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: As the trial is blinded neither the participants or the researchers will know which group the participants has been allocated to. In order to maintain the blind participants will take two tablets once daily for simvastatin. Group one will receive one 20mg tablet of simvastatin and one placebo table, group two will receive two 20 mg tablets of simvastatin and group three will receive two placebo tablets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simvastatin 20 mg + Rifaximin 400 mg (group 1) (Experimental): Simvastatin 20 mg/day and rifaximin 400 mg/8 hours orally for 12 weeks
  Interventions: Drug: Simvastatin 20 mg; Drug: Rifaximin 400 mg
- Simvastatin 40 mg + Rifaximin 400 mg (group 2) (Experimental): Simvastatin 40 mg/day and rifaximin 400 mg/8 hours orally for 12 weeks
  Interventions: Drug: Simvastatin 40mg; Drug: Rifaximin 400 mg
- Placebo of Simvastatin + Placebo of Rifaximin (group 3) (Placebo Comparator): Placebo simvastatin and placebo rifaximin orally for 12 weeks
  Interventions: Other: Placebo of Simvastatin; Other: Placebo of Rifaximin

INTERVENTIONS:
Drug: Simvastatin 20 mg — Simvastatin 20 mg/day for 12 weeks (Group 1)
  Arms: Simvastatin 20 mg + Rifaximin 400 mg (group 1)
Drug: Simvastatin 40mg — Simvastatin 40 mg/day for 12 weeks (Group 2)
  Arms: Simvastatin 40 mg + Rifaximin 400 mg (group 2)
Drug: Rifaximin 400 mg — Rifaximin 400 mg/8 hours for 12 weeks (Group 1 and 2)
  Arms: Simvastatin 20 mg + Rifaximin 400 mg (group 1); Simvastatin 40 mg + Rifaximin 400 mg (group 2)
Other: Placebo of Simvastatin — Placebo of Simvastatin for 12 weeks (Group 3)
  Arms: Placebo of Simvastatin + Placebo of Rifaximin (group 3)
Other: Placebo of Rifaximin — Placebo of Rifaximin for 12 weeks (Group 3)
  Arms: Placebo of Simvastatin + Placebo of Rifaximin (group 3)

SUMMARY:
The main purpose of this study is to investigate whether the combination of two different drugs, simvastatin and rifaximin, is safe in the treatment of patients with decompensated cirrhosis.

The secondary purpose is to see if this combination results in an improvement in inflammation markers in patients with cirrhosis and in an improvement in analytic parameters of progression of liver disease.

DETAILED DESCRIPTION:
Cirrhosis is the final stage of liver diseases, and currently, there is no effective treatment, with liver transplantation being the only curative solution in selected patients. As the number of donor organs for liver transplantation is limited and criteria for transplantation are strict, the current management of cirrhosis consists of treating its complications.

However, there is no effective therapy that prevents or cures the disease itself.

Rifaximin is an antibiotic that acts in the gastrointestinal tract. It is poorly absorbed to the general circulation and has low toxicity and good tolerability. Itis currently approved for use in patients with cirrhosis to prevent recurrent hepatic encephalopathy. Rifaximin decreases the transit of bacteria and bacterial products from the gut to the general circulation, preventing the chronic inflammation that takes place in cirrhotic patients.

Recent investigations have shown that simvastatin, a drug which is widely used to treat high cholesterol levels for the prevention of cardiovascular diseases, may have beneficial effects in patients with cirrhosis by preventing the progression of the disease and its complications. Although in the past decades there was a concern about its use in patients with liver disease due to its rare adverse effects (liver and muscle toxicity), recent clinical trials have shown that it can be safely used in patients with cirrhosis.

LIVERHOPE_SAFETY clinical trial have been designed to investigate whether the combination of these two drugs is safe in patients with cirrhosis, and also if it has potential beneficial effects in decreasing inflammation and improving analytical markers of progression of liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Cirrhosis defined by standard clinical criteria and ultrasonographic findings and/or histology. Cirrhosis of any etiology may be included. Patients with cirrhosis of autoimmune etiology on treatment with corticosteroids must be on stable corticosteroid dose for ≥3-month period before study inclusion.
* Child Pugh B/C patients (from 7 to 12 points).
* Women of child-bearing potential must have a negative pregnancy test in urine before the inclusion of the study and agree to use highly effective contraceptive methods (combined oral pill, injectable or implanted contraceptive, intrauterine device / intrauterine hormone-releasing system) during the study.

Exclusion Criteria:

* Patients on treatment with statins or rifaximin one month before study inclusion.
* Patients on the waiting list for liver transplantation.
* Patients with acute-on-chronic liver failure according to the criteria published by Moreau et al.
* Serum creatinine ≥2 mg/dL.
* Serum bilirubin>5 mg/dL.
* INR ≥2.5.
* Patients with CK elevation of 50% or more above the upper limit of normal at study inclusion.
* Bacterial infection within 15 days before study inclusion.
* Gastrointestinal bleeding within 15 days before study inclusion.
* Current overt hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy.
* HIV infection.
* Hepatocellular carcinoma outside Milan criteria, defined as a single nodule ≤5 cm or a maximum of 3 nodules with none >3 cm.
* Patients on antiviral therapy for HCV or those who have received it within the last 6 months.
* Patients with previous history of myopathy.
* Patients on treatment with potent inhibitors of CYP3A4 enzyme (See section 5.2: Concomitant, nonpermitted and permitted medication)
* Patients on treatment with drugs with potential interactions with simvastatin
* Patients with a history of significant extrahepatic disease with impaired short-term prognosis, including congestive heart failure New York Heart Association Grade III/IV, COPD GOLD >2, chronic kidney disease with serum creatinine >2mg/dL or under renal replacement therapy.
* Patients with current extrahepatic malignancies including solid tumours and hematologic disorders.
* Patients with previous history or increased risk of intestinal obstruction.
* Pregnancy or breastfeeding.
* Patients included in other clinical trials in the previous month.
* Patients with active alcohol consumption of more than 3 units per day.
* Patients with mental incapacity, language barrier, bad social support or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.
* Severe alcoholic hepatitis requiring corticosteroid therapy (Maddrey's Discriminant function ≥ 32 and/or ABIC score > 6.7).
* Refusal to give informed consent.
* Patients with contraindications for statins or rifaximin.
* Known hypersensitivity to rifaxamin (or rifamycin derivatives) or to simvastatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in transaminases during the treatment period, to evaluate treatment-related toxicity. | Week 12
  This quantitative analysis will consist of liver toxicity assessed by the development of liver injury defined as 3-fold increase in serum transaminases to a final value at least 3 times the upper normal limit
Change from baseline in alkaline phosphatase during the treatment period, to evaluate treatment-related toxicity. | Week 12
  This quantitative analysis will consist of liver toxicity assessed by the development of liver injury defined as 2-fold increase in serum levels of alkaline phosphatase with respect to baseline value to a final value at least 2 times the upper normal limit
Change from baseline in creatine kinase during the treatment period, to evaluate treatment-related toxicity. | Week 12
  This quantitative analysis will consist of muscle toxicity defined as 5-fold increase in creatine kinase (CK) levels during treatment

SECONDARY OUTCOMES:
Appearance of muscle toxicity at weeks 2, 4, 6, 8, 10 and 12 as defined using a specific statin-associated myopathy questionnaire | Weeks 2, 4, 6, 8, 10 and 12
Changes from baseline in plasma renin concentration levels at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in serum aldosterone levels at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in plasma norepinephrine levels at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in plasma copeptin levels at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, VCAM-1 and ICAM-1 | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, VEGF-A | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, Fractalkine | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, MIP-1α | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, Eotaxin | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, IP-10 | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, RANTES | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, GM-CSF | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, IL-1β, IL-2, IL-6 and IL-8 | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, MCP-1 | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, oxidized form of albumin | Weeks 2, 4, 8 and 12
Changes from baseline of plasma cytokine levels including, but not limited to, HNA2 | Weeks 2, 4, 8 and 12
Changes from baseline in plasma biomarker FABP4 at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in plasma biomarker CD-163 at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in urine biomarker NGAL at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in urine biomarker IL-18 at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in urine biomarker MCP-1 at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in urine biomarker osteopontin at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes from baseline in urine biomarker albumin at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Changes in blood levels of bacterial DNA or bacterial products at weeks 2, 4, 8 and 12. | Weeks 2, 4, 8 and 12
Number of patients with genetic polymorphisms of statins membrane transporter OATPB1 in patients developing treatment-related toxicity (defined as the primary endpoint of the study). | Week 12
Proportion of patients with treatment-related serious adverse events during the study period. | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, MD, Study Chair — Hospital Clinic of Barcelona
Locations (9):
- Beajuon Hospital, Clichy, Paris, France
- Universitatsklinikum Bonn, Bonn, Germany
- Italy (3):
  - Bologna University Hospital, Bologna
  - Padova University Hospital, Padua
  - San Giovanni Battista Hospital, Torino
- Academic Medical Centre, Amsterdam, Netherlands
- Spain (2):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pose E, Napoleone L, Amin A, Campion D, Jimenez C, Piano S, Roux O, Uschner FE, de Wit K, Zaccherini G, Alessandria C, Angeli P, Bernardi M, Beuers U, Caraceni P, Durand F, Mookerjee RP, Trebicka J, Vargas V, Andrade RJ, Carol M, Pich J, Ferrero J, Domenech G, Llopis M, Torres F, Kamath PS, Abraldes JG, Sola E, Gines P. Safety of two different doses of simvastatin plus rifaximin in decompensated cirrhosis (LIVERHOPE-SAFETY): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Gastroenterol Hepatol. 2020 Jan;5(1):31-41. doi: 10.1016/S2468-1253(19)30320-6. Epub 2019 Oct 10. PMID 31607677